CLINICAL TRIAL: NCT02559713
Title: An Open-Label, Multicenter and Open Enrollment Model, Postmarketing, Milk-Only Lactation Study to Assess Concentration of Vedolizumab in Breast Milk of Lactating Women With Active Ulcerative Colitis or Crohn's Disease Who Are Receiving Vedolizumab Therapeutically
Brief Title: Postmarketing Vedolizumab Milk-Only Lactation Study in Lactating Women With Active Ulcerative Colitis or Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4001; U1111-1171-5296 (Registry Identifier: WHO)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Colitis, Ulcerative; Crohn's Disease
Keywords: Lactation; Lactating Women; Vedolizumab; Colitis Ulcerative; Crohn's Disease; Crohn's
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Breast Feeding | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vedolizumab 300 milligram (mg) (Experimental): Vedolizumab 300 mg, IV infusion over 30-minutes, single dose on Day 1.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion
  Other Names: Entyvio; MLN0002

SUMMARY:
The purpose of this study is to assess the concentration of vedolizumab in breast milk of lactating women with active ulcerative colitis (UC) or Crohn's disease (CD) who are receiving vedolizumab therapeutically.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. This post-marketing milk-only lactation study will assess concentrations of vedolizumab in breast milk of lactating women with active UC or CD who are receiving vedolizumab therapeutically.

The study will enroll approximately 12 participants. All participants who received an established vedolizumab maintenance regimen or has completed induction therapy for the treatment of active UC or CD.

30-minute IV infusion of 300 mg vedolizumab. This multi-center trial will be conducted in the United States. The overall time to participate in this study is 3 months. Participants will make visits to clinic, study site or HCP office at Screening, Check-in (Day -1). Visits on Days 4, 8, 15, or 29 may be completed at the participant's home setting in the presence of a qualified nurse, or at a clinic, study site or other HCP office. The study exit/follow-up safety assessment will occur on Day 57(±3).

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. Signs and dates as written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is female and at least 18 years of age at the time of informed consent.
4. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent and throughout the duration of the study.
5. Is on established vedolizumab maintenance therapy and received at least 1 dose of 300 mg of vedolizumab IV postpartum or has completed vedolizumab induction therapy (300 mg of vedolizumab IV at Week 0, Week 2, and Week 6), which has been commenced by the participant's treating physician for the treatment of active UC or CD prior to enrolling in this study.
6. Has delivered a single, normal term infant (at least 37 weeks' gestation) that is, a mother-infant pair is required.
7. Is at least 5 weeks postpartum by Day 1.
8. Lactation is well established, and the mother is exclusively breast feeding her infant (or not providing more than 1 supplemental bottle of formula/day) when enrolled in the study.
9. Participant has independently decided to be treated with vedolizumab or to breastfeed prior to providing consent to participate in this study.
10. Plans to continue breastfeeding at least throughout the duration of this study.
11. Agrees to use only the emollient or nipple cream recommended by the investigator for use during the sampling period.

Exclusion Criteria:

1. Has received any investigational compound or approved biologic or biosimilar agent, except for vedolizumab within 60 days prior to enrollment in the study.
2. Within 30 days prior to enrollment, the participant has received any of the following for the treatment of underlying disease:

   * Nonbiologic therapies [example (eg), cyclosporine], other than those listed in the protocol.
   * An approved nonbiologic therapy in an investigational protocol.
3. Has received any live vaccinations within 30 days prior to vedolizumab administration.
4. Has clinically significant infection (eg, pneumonia, pyelonephritis) or chronic infection within 30 days prior to enrollment.
5. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
6. Has evidence of unstable or uncontrolled, clinically significant cardiovascular, central nervous system, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic or other medical disorder, including serious allergy, asthma, hypoxemia, hypertension, seizures or allergic skin rash that, in the opinion of the investigator, would confound the study results or compromise participant safety. Additionally, if there is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking vedolizumab, or a similar drug that might interfere with the conduct of the study.
7. Had any surgical procedure requiring general anesthesia within 30 days prior to enrollment or is planning to undergo major surgery during the study period.
8. Has any history of malignancy, except for the following: (a) adequately treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to enrollment; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to enrollment. Participants with remote history of malignancy (eg, greater than (>) 10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to enrollment.
9. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
10. Has a positive progressive multifocal leukoencephalopathy subjective symptom checklist at screening.
11. Has a current or recent history (within 1 year prior to enrollment) of alcohol dependence or illicit drug use.
12. Has active psychiatric problems that, in the investigator's opinion, may interfere with compliance with the study procedures.
13. Is unable to participate in all the study visits or comply with study procedures.
14. Has history of breast implants, breast augmentation, or breast reduction surgery.
15. Has a prior history of difficulty establishing lactation.
16. Has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table.
17. Has donated or lost 450 milliliters or more of her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to Day 1.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lactating women with a diagnosis of active ulcerative colitis (UC) or Crohn's disease (CD) being treated with vedolizumab were enrolled.
Enrollment: 11 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (7):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - Feinberg School of Medicine Northwestern University, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Atlantic Health System, Morristown, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Sun W, Fennimore B, Beaulieu DB, Arsenescu R, Stein AC, Chen J, Lin T, McKnight S, Kadali H, Rosario M, Lirio RA. Vedolizumab Concentrations in Breast Milk: Results from a Prospective, Postmarketing, Milk-Only Lactation Study in Nursing Mothers with Inflammatory Bowel Disease. Clin Pharmacokinet. 2021 Jun;60(6):811-818. doi: 10.1007/s40262-021-00985-4. Epub 2021 Feb 5. PMID 33544318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 29 November 2017 to 22 February 2019.
Pre-assignment Details: Lactating women with a diagnosis of active ulcerative colitis (UC) or Crohn's disease (CD) being treated with vedolizumab were enrolled to receive a single vedolizumab 300 milligrams (mg) dose intravenous (IV).
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, IV infusion over 30-minutes, single dose on Day 1.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg
Started | 11
Safety Set | 11
Pharmacokinetic Set | 11
Completed | 10
Not Completed | 1
Not completed — Pretreatment Event/ Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received any amount of vedolizumab in this study.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 158.9 (7.12)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 62.72 (15.924)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/[height (m)^2]
  kg/m^2 | 24.78 (5.534)
Smoking Status [Count of Participants; unit: Participants]
  Never Smoked | 11
Alcohol Status [Count of Participants; unit: Participants]
  Has Never Drunk | 5
  Current Drinker | 4
  Ex-drinker | 2
Female Reproductive Status [Count of Participants; unit: Participants]
  Surgically Sterile | 1
  Female of Childbearing Potential | 10
Breastfed in the Past [Count of Participants; unit: Participants]
  Yes | 6
  No | 5
Problems with Producing Breast Milk for Previously Breastfed Infants [Count of Participants; unit: Participants] — Population: Only participants who answered yes to the leading question of 'breastfed in the past' were analyzed.
  Participants
    number analyzed (Participants) | 6
    No | 6
Fail to Thrive for Previously Breastfed Infants [Count of Participants; unit: Participants] — Population: Only participants who answered yes to the leading question of 'breastfed in the past' were analyzed.
  Participants
    number analyzed (Participants) | 6
    No | 6

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Vedolizumab in Breast Milk at Predose on Day 1
Description: Milk from each breast was completely emptied using an electric milk pump at the specified time point for the determination of vedolizumab concentrations in the milk. Analysis of vedolizumab concentration from the pooled milk sample was done by enzyme-linked immunosorbent assay (ELISA). Participants were categorized as per their past vedolizumab regimens, received prior to Day 1: vedolizumab every 4 weeks (Q4W), vedolizumab every 6 weeks (Q6W), vedolizumab every 8 weeks (Q8W).
Time Frame: Day 1 (60 minutes prior to the start of infusion)
Population: Pharmacokinetic Set (PK) included all participants who were enrolled and received 1 dose of vedolizumab in the study and had at least 1 measurable milk concentration. Number analyzed is the number of participants who received specific vedolizumab regimen prior to Day 1.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 11
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.1350 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 9
  Q8W | 0.03161 (0.024327)

2. Primary Outcome: Concentration of Vedolizumab in Breast Milk at 1 Hour After the End of Infusion on Day 1
Description: Milk from each breast was completely emptied using an electric milk pump at the specified time point for the determination of vedolizumab concentrations in the milk. Analysis of vedolizumab concentration from the pooled milk sample was done by ELISA. Participants were categorized as per their past vedolizumab regimens, received prior to Day 1: vedolizumab every 4 weeks (Q4W), vedolizumab every 6 weeks (Q6W), vedolizumab every 8 weeks (Q8W).
Time Frame: Day 1 (approximately 60 minutes after the end of infusion)
Population: PK Set included all participants who were enrolled and received 1 dose of vedolizumab in the study and had at least 1 measurable milk concentration at the given timepoint. Number analyzed is the number of participants who received specific vedolizumab regimen prior to Day 1.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 10
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.1490 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 8
  Q8W | 0.03756 (0.025572)

3. Primary Outcome: Concentration of Vedolizumab in Breast Milk on Day 4
Description: Milk from each breast was completely emptied using an electric milk pump at the specified time point for the determination of vedolizumab concentrations in the milk. Analysis of vedolizumab concentration from the pooled milk sample was done by ELISA. Participants unable to return to the clinic could have their milk samples collected at home by a qualified and trained homecare nurse. Participants were categorized as per their past vedolizumab regimens, received prior to Day 1: vedolizumab every 4 weeks (Q4W), vedolizumab every 6 weeks (Q6W), vedolizumab every 8 weeks (Q8W).
Time Frame: Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 10
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.3050 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0.1650 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 8
  Q8W | 0.2634 (0.14840)

4. Primary Outcome: Concentration of Vedolizumab in Breast Milk on Day 8
Description: as for outcome 3
Time Frame: Day 8
Population: PK Set included all participants who were enrolled and received 1 dose of vedolizumab in the study and had at least 1 measurable milk concentration. Number analyzed is the number of participants who received specific vedolizumab regimen prior to Day 1.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 11
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.3050 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0.1410 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 9
  Q8W | 0.2113 (0.10299)

5. Primary Outcome: Concentration of Vedolizumab in Breast Milk on Day 15
Description: as for outcome 3
Time Frame: Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 11
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.2280 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0.1270 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 9
  Q8W | 0.1708 (0.069017)

6. Primary Outcome: Concentration of Vedolizumab in Breast Milk on Day 29
Description: as for outcome 3
Time Frame: Day 29
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 11
ug/mL
  Q4W: number analyzed (Participants) | 1
  Q4W | 0.1560 (NA) — Standard deviation was not estimable for one participant.
  Q6W: number analyzed (Participants) | 1
  Q6W | 0.06860 (NA) — Standard deviation was not estimable for one participant.
  Q8W: number analyzed (Participants) | 9
  Q8W | 0.1039 (0.040445)

7. Primary Outcome: Concentration of Vedolizumab in Breast Milk on Day 57
Description: Milk from each breast was completely emptied using an electric milk pump at the specified time point for the determination of vedolizumab concentrations in the milk in participants with analysis of vedolizumab concentration from the pooled milk sample was done by ELISA.
Time Frame: Day 57
Population: Participants from PK Set, included all participants who were enrolled and received 1 dose of vedolizumab in study and had at least 1 measurable milk concentration, who received vedolizumab Q8W regimen prior to Day 1 with data available for this outcome measure were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 7
ug/mL | 0.04673 (0.020966)

ADVERSE EVENTS:
Time Frame: First dose of study drug in this study to study exit (Up to Day 57)
Arm/Group | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=11)
Colitis ulcerative (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=11)
Crohn's disease (Gastrointestinal disorders) | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1
Paronychia (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT02559713/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02559713/SAP_001.pdf